CLINICAL TRIAL: NCT01007955
Title: Assessment of Insulin Resistance, Non-Alcoholic Fatty Liver Disease, Predictors of Cardiovascular Morbidity, and Subcutaneous Adipose and Visceral Adipose Gene Expression in Patients Undergoing Gastric Bypass: Development of a New Paradigm in Defining "Morbid Obesity" and in the Application of Bariatric Surgery
Brief Title: Assessment of Insulin Resistance, NAFLD, Predictors of CV Morbidity, and Subcutaneous Adipose and Visceral Adipose Gene Expression in Patients Undergoing Gastric Bypass Surgery
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Richard Perugini, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: H-12082
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Morbid Obesity; Insulin Resistance; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Obesity, Morbid; Insulin Resistance; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subcutaneous and visceral adipose tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severely Obese: Severely obese individuals scheduled to undergo gastric bypass surgery

SUMMARY:
The purpose of this research is to further study the effect weight loss after gastric bypass surgery has on the heart and blood pressure and on how the body uses or metabolizes the sugars, fats and proteins we eat. Additionally, the researchers want to study fat tissue for gene patterns which may be responsible for where we carry fat on our bodies, as well as look carefully at a possible link between adipose tissue and insulin resistance. The researchers also want to evaluate the liver for the presence of fatty liver, which is common in people with obesity and is associated with insulin resistance, as well as study the liver for gene patterns which may be associated with non-alcoholic liver disease.

Evaluating cardiovascular function and endocrine function before and after gastric bypass surgery, as well as studying adipose and liver tissue may help us understand the link between obesity, insulin resistance, fatty liver disease, high blood pressure and health problems such as diabetes and heart disease. Consequently, this may help in the future by identifying those who will benefit most from gastric bypass surgery.

DETAILED DESCRIPTION:
Obesity is associated with insulin resistance and diabetes. Since both of these conditions have been implicated in cardiovascular complications, this association may explain obesity related illnesses and deaths. Gastric bypass is considered the "gold standard" surgical weightloss procedure and has been demonstrated to cure diabetes and insulin resistance. Some severely obese patients, however, have normal insulin-glucose metabolism. The differences in metabolic healthy in severely obese individuals has not been fully recognized or understood. This research will study insulin-glucose metabolism in a population of severely obese individuals undergoing gastric bypass. This investigation is based on the following hypotheses:

1. Severely obese individuals can be categorized by degree to which insulin-glucose homeostasis is impaired.
2. The degree of insulin resistance correlates with risk for cardiovascular disease. Weight loss in obese individuals with insulin resistance, will correlate with improvement in parameters associated with cardiovascular disease. Obese individuals with better insulin sensitivity will not have a high risk for cardiovascular disease and therefore will not experience this risk reduction in cardiovascular disease.
3. Insulin resistance is a consequence of pathological storage of excess energy intake; therefore, individuals who are insulin resistant and obese will differ from individuals who are obese, but not insulin resistant with regards to gene expression in subcutaneous adipose tissue and visceral adipose tissue.

Subjects will be studied for evidence of end organ dysfunction and predictors of morbidity and mortality preoperatively and postoperatively. Additionally, gene expression in the subcutaneous and visceral adipose depots of subjects will be studied

ELIGIBILITY:
Inclusion Criteria:

* Morbid Obesity
* Scheduled to undergo gastric bypass surgery

Exclusion Criteria:

* Pregnancy (would not be candidate for surgery)
* Nursing (would not be candidate for surgery)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely obese patients undergoing gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2006-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Improvement of insulin resistance and/or diabetes | Two weeks postoperatively, Six months postoperatively, One year postoperatively

SECONDARY OUTCOMES:
Improvement of cardiovascular risk factors | Two weeks postoperatively, Six months postoperatively, One year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States